CLINICAL TRIAL: NCT02162823
Title: Prospective Populationbased Study on Pancreatic Cancer in Stockholm- Mutation Profiling Characteristics, Biobanking and Risk Factors.
Brief Title: Clinical Trial of Pancreatic Cancer in Stockholm.
Acronym: SPP
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Matthias Löhr, Professor, Karolinska University Hospital
Other Study IDs: 2006/1089-31/4; 2006/1089-31/4 (Other: Swedish Ethic committee)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Cancer
Keywords: The MeSH name is Carcinoma, Pancreatic Ductal
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Germline DNA and tumour DNA (PDAC patients). Saliva and urine (DNA).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic cancer: Patients with pancreatic cancer and age&sex-matched controls without any cancer from a distinct population area (district of Stockholm). Patients with pancreatic cancer will be subjected to pancreatic surgery
  Interventions: Procedure: Pancreatic Surgery

INTERVENTIONS:
Procedure: Pancreatic Surgery — Surgical removal of the pancreatic tumour (cancer) in the intervention group
  Other Names: Pancreatic head resection; Whipple procedure; Pancreatic resection

SUMMARY:
SPP study includes incidence cases of pancreatic cancer in the Stockholm county region from 2007 to 2014. The purpose of SPP study is to estimate relative risk of pancreatic cancer in relation to snuff dipping, overweight/obesity, individual food items, food groups, dietary pattern and various nutrients; to estimate relative risk of pancreatic cancer in relation to exposure to nitrosamines, either endogenously or exogenously; to estimate relative risk of pancreatic cancer in relation to oral health and H.pylori infection and their interaction with ABO blood type; to estimation relative risk of pancreatic cancer in relation to hepatitis B or hepatitis C infection; to estimate relative risk of pancreatic cancer in relation to some genetic polymorphisms, either functional or being suggested in GWAS study; to estimate mutation profile in pancreatic cancer cases, and its correlation with environmental exposures, and the impacts on survival periods in pancreatic cancer patients.

The MeSH name is Carcinoma, Pancreatic Ductal

DETAILED DESCRIPTION:
The SPP study is a prospective population-based case-control study. We include incident cases of pancreatic cancer in the Stockholm county region during 2008 to 2014. Controls are randomly selected from general population in the Stockholm region, and individually matched to cases by age and sex.

Cases selection. The criteria for cases selection including those are age less than 85 years, born in Sweden and presently living in the county of Stockholm. The cases of pancreatic cancer are first identified within the framework of the clinical healthcare system of the Stockholm County. Through a network, consisting of all surgical clinics and the only oncological clinic in the Stockholm county area, we were able to include a vast majority of cases diagnosed with radiological methods, he or she were asked to participate in the study. After informed consent is obtained from the patient, the study coordinator at the Karolinska University Hospital at Huddinge was notified. The coordinator will inform Statistics Sweden interviewer to interview the case patient. Further, after radiological diagnosis of pancreatic cancer, we try to retrieve a tumor biopsy for every case. In total around 30% of the cases are surgically resected and of the remaining 70% of the patients treated with a palliative intention and among which more than 80% are biopsied using fine needle aspiration (the remaining 20% not biopsied for practical reasons such as clinical deterioration), thus resulting in a total proportion of patients in which tumor tissue is retained of close to 90%.

Control selection. The control persons (non-cancer patients) are randomly identified via the Statistics Sweden. For each case, a gender- and age-matched (same birth year) control person will be identified randomly from the general population of the Stockholm County.

Data collection. Through professional interviewers from the Statistics Sweden, interviews were conducted concerning environmental factors with both cases and control persons. As soon as the study coordinator identified a case of pancreatic cancer and the patient has accepted to participate, Statistics Sweden is contacted about this patient's identify and location. Professional interviewers, blinded to the research hypotheses of the study, will then contact and go to the patient at home, at the hospital or wherever the patient is and perform the interview which is calculated to take around 1 hour and 15 minutes. The questionnaire contains items concerning demographics, socioeconomic factors, physical activity, height and weight history, tobacco and snuff use, dental health, earlier and concomitant diseases and medication history. A structured food frequency questionnaire, a modified version of a previously evaluated questionnaire, including 63 food and beverage items of interest, are used to evaluate dietary habits 20 years prior to interview.

Once a case has been identified, a set of up to 5 controls (same sex and birth year) from Stockholm general population will be selected by the Statistics Sweden. The control persons in the list are contacted by order, until a control person agrees to participate in our study. The interviewers will perform the interview in exactly the same way for the cases.

For each case and control, if they agree, 20 ml of blood are collected. The samples are separated into serum and cells (red and white together) and aliquot into 4 separate serum (for subsequent protein analysis) samples and 2 cell samples after Ficoll gradient (for subsequent DNA and RNA analysis) and immediately frozen to -80°C. Control persons that decline leaving a blood sample are instead offered to leave a saliva sample, from which DNA can be extracted and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* pancreatic cancer patients that aged less than 85 years old born in Sweden living in Stockholm
* written informed consent

Exclusion Criteria:

* pancreatic cancer older than 85 years
* pancratic cancer younger than 18 years
* not willing to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population based cohort of all patients with pancreatic cancer within the district of Stockholm and age and gender matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2007-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Survival | 5 years

SECONDARY OUTCOMES:
Factors influencing survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Löhr, Professor, Principal Investigator — Karolinska University Hospital; Magnus Nilsson, ass prof, Study Director — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Gastrocentrum, Stockholm, Sweden

REFERENCES:
- [Result] Yu J, Song H, Ekheden I, Lohr M, Ploner A, Ye W. Gastric Mucosal Abnormality and Risk of Pancreatic Cancer: A Population-Based Gastric Biopsy Cohort Study in Sweden. Cancer Epidemiol Biomarkers Prev. 2021 Nov;30(11):2088-2095. doi: 10.1158/1055-9965.EPI-21-0580. Epub 2021 Sep 8. PMID 34497088
- [Result] Molina-Montes E, Van Hoogstraten L, Gomez-Rubio P, Lohr M, Sharp L, Molero X, Marquez M, Michalski CW, Farre A, Perea J, O'Rorke M, Greenhalf W, Ilzarbe L, Tardon A, Gress TM, Barbera VM, Crnogorac-Jurcevic T, Munoz-Bellvis L, Dominguez-Munoz E, Balsells J, Costello E, Iglesias M, Kleeff J, Kong B, Mora J, O'Driscoll D, Poves I, Scarpa A, Yu J, Ye W, Hidalgo M, Carrato A, Lawlor R, Real FX, Malats N; PanGenEU Study Investigators. Pancreatic Cancer Risk in Relation to Lifetime Smoking Patterns, Tobacco Type, and Dose-Response Relationships. Cancer Epidemiol Biomarkers Prev. 2020 May;29(5):1009-1018. doi: 10.1158/1055-9965.EPI-19-1027. Epub 2020 Feb 12. PMID 32051190
- [Result] Yu J, Ploner A, Kordes M, Lohr M, Nilsson M, de Maturana MEL, Estudillo L, Renz H, Carrato A, Molero X, Real FX, Malats N, Ye W. Plasma protein biomarkers for early detection of pancreatic ductal adenocarcinoma. Int J Cancer. 2021 Apr 15;148(8):2048-2058. doi: 10.1002/ijc.33464. Epub 2021 Jan 15. PMID 33411965
- [Result] Molina-Montes E, Coscia C, Gomez-Rubio P, Fernandez A, Boenink R, Rava M, Marquez M, Molero X, Lohr M, Sharp L, Michalski CW, Farre A, Perea J, O'Rorke M, Greenhalf W, Iglesias M, Tardon A, Gress TM, Barbera VM, Crnogorac-Jurcevic T, Munoz-Bellvis L, Dominguez-Munoz JE, Renz H, Balcells J, Costello E, Ilzarbe L, Kleeff J, Kong B, Mora J, O'Driscoll D, Poves I, Scarpa A, Yu J, Hidalgo M, Lawlor RT, Ye W, Carrato A, Real FX, Malats N; PanGenEU Study Investigators. Deciphering the complex interplay between pancreatic cancer, diabetes mellitus subtypes and obesity/BMI through causal inference and mediation analyses. Gut. 2021 Feb;70(2):319-329. doi: 10.1136/gutjnl-2019-319990. Epub 2020 May 14. PMID 32409590